CLINICAL TRIAL: NCT00805948
Title: Descending Thoracic Aortic Aneurysm Endovascular Repair Post-approval Study (THRIVE)
Brief Title: Post-Approval Clinical Study of the Talent Thoracic Stent Graft to Treat Thoracic Aortic Aneurysms (THRIVE)
Acronym: THRIVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study device discontinued & insufficient sample size for statistical results.
Sponsor: Medtronic Cardiovascular (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Investigational Plan #109
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Thoracic Aortic Aneurysms
Keywords: thoracic aneurysm; thoracic aortic aneurysms; Thoracic Endovascular Aneurysm Repair (TEVAR); Talent Thoracic Stent Graft
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DeNovo (Experimental): Prospectively enrolled subjects treated with the Talent Thoracic Stent Graft System following U.S. market approval of the device.
  Interventions: Device: Talent Thoracic Stent Graft System
- Valor (No Intervention): Historical control arm, consisting of 195 subjects from the VALOR Test Group (PMA P070007) that were followed for 5 years per the VALOR protocol. The data from these subjects will be combined with the data from the subjects implanted after commercial release (DeNovo) to comprise the final analysis cohort for the THRIVE Study

INTERVENTIONS:
Device: Talent Thoracic Stent Graft System — endovascular repair of descending thoracic aortic aneurysms using the Talent Thoracic Stent Graft System.
  Arms: DeNovo

SUMMARY:
The purpose of this study is to evaluate the long-term safety and effectiveness of the Talent Thoracic Stent Graft System for treatment of descending thoracic aneurysms (DTA)following U.S. market approval.

DETAILED DESCRIPTION:
A descending thoracic aneurysm is a bulge in the aorta. The aorta is a large blood vessel that carries blood away from your heart to organs in the rest of your body. Your aneurysm is caused by a weakening in the artery wall. If left untreated, this bulge may continue to grow larger and may ultimately rupture (break open) or extend in size to seriously affect other major arteries in the area. In this clinical study the Talent Thoracic Stent Graft will be placed inside your aorta to block the weakened part of the artery wall from the circulatory system.

Medtronic Vascular submitted a Pre-Market Application (PMA P070007) to the FDA on February 28, 2007, and received market approval for the Talent Stent Graft System on June 5, 2008. As a condition of approval, the FDA has requested a post-market trial. In collaboration with the FDA, Medtronic has designed a post-approval study to document the long-term performance of the Talent Stent Graft System under post market conditions.

This study will examine the post-market performance of the Talent Thoracic Stent Graft System. This study is a prospective, non-randomized five-year trial. Originally, a total of 451 subjects were going to be analyzed. That group consisted of 195 enrolled subjects from the VALOR Test Group of the Talent Thoracic PMA Submission, and 256 planned "de novo" subjects enrolled after the PMA approval. However, Medtronic discontinued manufacturing of the study device for US commercialization, and as a result, enrollment was terminated in May 2014, when it was determined that no more proximal devices were available either in inventory or at the sites. A total of 349 subjects will be analyzed, based on 195 VALOR Test Group subjects and 154 "de novo" subjects.

Update as of Aug 2017: Medtronic Vascular, Inc. discontinued manufacture of the Talent Thoracic Stet Graft System on 31-Jul-2012, and the final device expired in July 2014 (based on the two-year shelf life). Enrollment for De Novo subjects ended in May 2014, as there were no more proximal main devices available either in inventory or at the investigational sites. This resulted in a total of 349 subjects to be analyzed in this final report: the 195 VALOR subjects and 154 of the planned 256 De Novo subjects. Because of that, statistical results would have been inconclusive, so Medtronic decided to terminate the study and received FDA approval for early termination in April 2016.

It is important to emphasize that THRIVE subjects will continue to be followed-up annually per standard of care and standard post-market surveillance program applies to them (e.g. device complaints will continue to be reported via the MDR (Medical Device Reporting) system.)

ELIGIBILITY:
Inclusion Criteria: appropriate anatomy for elective repair of the descending thoracic aortic aneurysm

* iliac/femoral access vessel morphology that is compatible with vascular access techniques, devices, and or accessories
* non-aneurysmal aortic diameter in the range of 18-42mm; and
* non-aneurysmal aortic proximal and distal neck lengths equal to or greater than 20mm
* subject has a Descending Fusiform Thoracic Aneurysm = to or greater than 5cm in diameter OR is = to or greater than 2 times the diameter of the non-aneurysmal thoracic aorta and/or saccular aneurysms/penetrating ulcers
* Signed patient informed consent

Exclusion Criteria:

* Less than 18 yrs old
* pregnant
* unable to comply w/follow-up
* participating in other drug or device trials;
* Subject has a co-morbidity causing expected survival to be less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam W Beck, MD, Principal Investigator — University of Florida
Locations (26):
- United States (26):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Harbor-UCLA, Torrance, California
  - Washington Hospital D.C., Washington D.C., District of Columbia
  - U Florida at Shands Hospital, Gainesville, Florida
  - Osceola Regional Med Ctr, Kissimmee, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern MH, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - St. Vincent Heart Center, Indianapolis, Indiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Albany Medical Center, Albany, New York
  - Northwell Health Inc, Great Neck, New York
  - Duke University Medical Center, Durham, North Carolina
  - Riverside Methodist Hospital, Columbus, Ohio
  - University of Toledo Med Ctr, Toledo, Ohio
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Pinnacle Health, Wormleysburg, Pennsylvania
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Tennova Physicians Regional Medical Center, Powell, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - The Heart Hospital/Baylor Plano, Plano, Texas
  - Sentara Norfolk General Vascular & Transplant Specialists, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - Providence Sacred Heart, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- De Novo Group: 154 of the planned 256 prospectively enrolled De Novo subjects treated with the Talent Thoracic Stent Graft System following U.S. market approval of the device.
- Valor Test Group: 195 subjects from the Valor Test Group (PMA P070007) that were followed for 5 years per the VALOR protocol.
Period: Overall Study
Arm/Group | De Novo Group | Valor Test Group
Started | 154 | 195
Completed | 86 | 99
Not Completed | 68 | 96

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | De Novo Group | Valor Test Group | Total
Number analyzed (Participants) | 154 | 195 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (11.4) | 70.2 (11.1) | 70.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 80 | 154
  Male | 80 | 115 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 145 | 190 | 335
  Unknown or Not Reported | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian/Native Hawaiian or Pacific Islander | 4 | 2 | 6
  Black or African American | 20 | 25 | 45
  White | 127 | 162 | 289
  Other | 3 | 1 | 4
  Unknown or Not Available | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Aneurysm-related Mortality at 5 Years
Description: For all THRIVE subjects, Aneurysm-Related Mortality (ARM) is defined as: Death from rupture of the thoracic aortic aneurysm or from any procedure intended to treat the Descending Thoracic Aneurysm (DTA - fusiform aneurysms and saccular aneurysms/penetrating ulcers) as determined by an independent Clinical Events Committee (CEC). If a death occurred within 30 days of any procedure intended to treat the DTA, then it is presumed to be aneurysm related, unless there is evidence to the contrary.
Time Frame: 5 years
Population: All participants were combined for analysis as a single arm, as pre-specified in the protocol. Subjects are censored because their last follow-up has not reached the end of the time interval or because they withdraw, are lost to follow-up or die from a non-aneurysm related cause.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Subjects: All Subjects (349) is comprised of 195 subjects from the VALOR Test Group (PMA P070007) and 154 of the planned 256 De Novo subjects.
Arm/Group | All Subjects
Number analyzed (Participants) | 349
Percentage of participants | 92 [88 to 95]

2. Other Pre Specified Outcome: All-Cause Mortality
Description: Number of subjects who died during that interval or who were followed at least until the lower endpoint of the analysis window.
Time Frame: 1, 12, 24, 36, 48 and 60 months
Population: Based on all Intent to Treat (ITT) subjects.
Measure: Number; unit: Participants
Arm/Group | De Novo Group | Valor Test Group
Number analyzed (Participants) | 154 | 195
Participants
  0-30 days | 5 | 4
  0 - 365 days | 17 | 31
  366 - 731 days | 18 | 11
  732 - 1096 days | 8 | 15
  1097 - 1461 days | 8 | 9
  1462 - 1826 days | 3 | 10

3. Other Pre Specified Outcome: Number of Participants With Conversion to Surgery
Description: Conversion from endovascular to open repair required at the time of the original procedure or at the time beyond the initial endovascular procedure (for the same lesion treated during the initial implantation of the Talent Thoracic Stent Graft)
Time Frame: 1, 12, 24, 36, 48 and 60 months
Population: Based on all Intent to Treat (ITT) subjects.
Measure: Number; unit: participants
Arm/Group | De Novo Group | Valor Test Group
Number analyzed (Participants) | 154 | 195
participants
  0-30 days | 1 | 0
  0-365 days | 2 | 1
  366-731 days | 0 | 1
  732-1096 days | 0 | 1
  1097-1461 days | 0 | 0
  1462-1826 days | 0 | 1

4. Other Pre Specified Outcome: Number of Participants With Aneurysm Rupture
Description: Rupture or perforation of the targeted aneurismal sac as detected by angiography, CT scan, or direct observation at surgery or autopsy.
Time Frame: 1, 12, 24, 36, 48 and 60 months
Population: Based on all Intent to Treat (ITT) subjects
Measure: Number; unit: participants
Arm/Group | De Novo Group | Valor Test Group
Number analyzed (Participants) | 154 | 195
participants
  0-30 days | 0 | 0
  0-365 days | 0 | 1
  366-731 days | 2 | 0
  732-1096 days | 1 | 2
  1097-1461 days | 0 | 0
  1462-1826 days | 0 | 2

ADVERSE EVENTS:
Time Frame: 5 years
Description: The 195 VALOR subjects completed follow-up on 16-Jun-2011 per VALOR protocol PMA P070007 (previously reported via G980116/S280). Due to limited access to this older study data, the AE terms couldn't be re-validated using MedDRA. Therefore, the AE terms of Valor subjects are posted as they were originally validated, using the Valor study-specific definitions.
  The 154 De Novo subjects were followed per the THRIVE protocol. The AE terms for De Novo subjects were validated using MedDRA 17.0.
Arm/Group | De Novo Group | Valor Test Group
All-Cause Mortality (participants affected / at risk) | 54/154 | 76/195
Serious Adverse Events (participants affected / at risk) | 83/154 | 178/195
Other Adverse Events (participants affected / at risk) | 0/154 | 0/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | De Novo Group (N=154) | Valor Test Group (N=195)
Aortic Valve Disease (Cardiac disorders) | 1 (1) | 0/0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0/0 (0)
Cardiac Arrest (Cardiac disorders) | 5 (5) | 0/0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0/0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0/0 (0)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0/0 (0)
Cardiopulmonary Failure (Cardiac disorders) | 2 (2) | 0/0 (0)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1) | 0/0 (0)
Myocardial Infarction (Cardiac disorders) | 4 (4) | 0/0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0/0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0/0 (0)
Intestinal Ischaemia (Gastrointestinal disorders) | 2 (2) | 0/0 (0)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0/0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0/0 (0)
Device Dislocation (General disorders) | 1 (1) | 0/0 (0)
Multi-Organ Failure (General disorders) | 1 (1) | 0/0 (0)
Stent-Graft Endoleak (General disorders) | 20 (23) | 0/0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0/0 (0)
Groin Infection (Infections and infestations) | 1 (1) | 0/0 (0)
Infection (Infections and infestations) | 1 (1) | 0/0 (0)
Infective Aneurysm (Infections and infestations) | 1 (1) | 0/0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 0/0 (0)
Sepsis (Infections and infestations) | 6 (6) | 0/0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0/0 (0)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 9 (9) | 0/0 (0)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (2) | 0/0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0/0 (0)
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0/0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0/0 (0)
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0/0 (0)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0/0 (0)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0/0 (0)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0/0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 3 (3) | 0/0 (0)
Cerebrovascular Accident (Nervous system disorders) | 7 (8) | 0/0 (0)
Paraparesis (Nervous system disorders) | 2 (2) | 0/0 (0)
Mental Status Changes (Psychiatric disorders) | 3 (3) | 0/0 (0)
Renal Failure (Renal and urinary disorders) | 11 (13) | 0/0 (0)
Renal Failure Acute (Renal and urinary disorders) | 2 (2) | 0/0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0/0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0/0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0/0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0/0 (0)
Diaphragmatic Paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/0 (0)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 0/0 (0)
Coronary Artery Bypass (Surgical and medical procedures) | 1 (1) | 0/0 (0)
Aneurysm (Vascular disorders) | 3 (3) | 0/0 (0)
Aneurysm Ruptured (Vascular disorders) | 1 (1) | 0/0 (0)
Aortic Aneurysm (Vascular disorders) | 3 (3) | 0/0 (0)
Aortic Aneurysm Rupture (Vascular disorders) | 1 (1) | 0/0 (0)
Aortic Dilatation (Vascular disorders) | 1 (1) | 0/0 (0)
Aortic Dissection (Vascular disorders) | 1 (1) | 0/0 (0)
Aortic Rupture (Vascular disorders) | 4 (4) | 0/0 (0)
Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0/0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0/0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0/0 (0)
Embolism (Vascular disorders) | 1 (1) | 0/0 (0)
Peripheral Artery Dissection (Vascular disorders) | 4 (4) | 0/0 (0)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0/0 (0)
Pulmonary complications (general) (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 61 (98)
Renal complications (general) (Renal and urinary disorders) | 0/0 (0) | 17 (22)
Cardiac and hemodynamic (general) (Cardiac disorders) | 0/0 (0) | 50 (64)
Cardiac Arrhythmia (Cardiac disorders) | 0/0 (0) | 16 (17)
Congestive heart failure (Cardiac disorders) | 0/0 (0) | 18 (23)
Myocardial infarction (Cardiac disorders) | 0/0 (0) | 12 (13)
Neurologic (general) (Nervous system disorders) | 0/0 (0) | 20 (22)
Paraplegia and paraparesis (Nervous system disorders) | 0/0 (0) | 13 (13)
Stroke (Nervous system disorders) | 0/0 (0) | 14 (15)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 0/0 (0) | 3 (3)
Gastrointestinal (general) (Gastrointestinal disorders) | 0/0 (0) | 32 (44)
Bowel obstruction (Gastrointestinal disorders) | 0/0 (0) | 3 (3)
Mesenteric ischemia (Gastrointestinal disorders) | 0/0 (0) | 3 (3)
Bleeding and hematogenic (Vascular disorders) | 0/0 (0) | 69 (92)
GI bleed (Gastrointestinal disorders) | 0/0 (0) | 12 (18)
Arterial (Vascular disorders) | 0/0 (0) | 50 (65)
Arterial embolism (Vascular disorders) | 0/0 (0) | 8 (9)
Arterial insertion trauma (General disorders) | 0/0 (0) | 10 (10)
TAA rupture (Vascular disorders) | 0/0 (0) | 5 (5)
Venous (Vascular disorders) | 0/0 (0) | 3 (3)
Graft endoleak (General disorders) | 0/0 (0) | 29 (36)
Graft migration (General disorders) | 0/0 (0) | 2 (2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 18 (21)
Infection (Infections and infestations) | 0/0 (0) | 22 (28)
Urologic (Renal and urinary disorders) | 0/0 (0) | 8 (8)
Other-Enlarged Lymph Nodes - Right (Blood and lymphatic system disorders) | 0/0 (0) | 1 (1)
Other - (L) Hip Dysplasia (Congenital, familial and genetic disorders) | 0/0 (0) | 1 (1)
Other - (L) Knee Replacement (Surgical and medical procedures) | 0/0 (0) | 1 (1)
Other - (R) Hip Fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Other - Acute Morphine Poisoning (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Other - Arthritis of Knee (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 1 (1)
Other - Auditory and Visual (Psychiatric disorders) | 0/0 (0) | 1 (1)
Other - Broken Hip (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 1 (1)
Other - Cervical Spine Fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Other - Cirrhosis (Hepatobiliary disorders) | 0/0 (0) | 1 (1)
Other - Degenerative Joint Disease (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 1 (1)
Other - Dizziness (Nervous system disorders) | 0/0 (0) | 1 (1)
Other - Fall - FX Hip (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Other - Fracture of Left Leg (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Other - Fractured Left Foot (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Other - Hernia (General disorders) | 0/0 (0) | 2 (2)
Other - Hip Fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Other - Hypercalcemia (Metabolism and nutrition disorders) | 0/0 (0) | 1 (1)
Other - Hypoalbuminemia/Malnutrition (Metabolism and nutrition disorders) | 0/0 (0) | 1 (1)
Other - Immature Fistula, Permacath (Surgical and medical procedures) | 0/0 (0) | 1 (1)
Other - Malnutrition (Metabolism and nutrition disorders) | 0/0 (0) | 2 (2)
Other - Osteoarthritis (L) Knee (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 1 (1)
Other - Osteoarthritis/(L) Total Knee (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 1 (1)
Other - Right Femur Fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Other - Splenic Rupture (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Other - Suicidal Ideation (Psychiatric disorders) | 0/0 (0) | 1 (1)
Other - Uterine Prolapse (Reproductive system and breast disorders) | 0/0 (0) | 1 (1)
Other - Weakness (General disorders) | 0/0 (0) | 1 (1)
Other - Anxiety (Psychiatric disorders) | 0/0 (0) | 1 (1)
Other - Back Pain (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 4 (5)
Other - Fever (General disorders) | 0/0 (0) | 4 (4)
Other - Fever (Infections and infestations) | 0/0 (0) | 1 (1) — Fungemia
Other - Pain (General disorders) | 0/0 (0) | 5 (5)
Other - Pain (General disorders) | 0/0 (0) | 1 (1) — Right groin
Other - Pain (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 1 (1) — Left side of neck, left arm and leg
Other - Pain (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 1 (1) — (L) calf pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes